CLINICAL TRIAL: NCT02723019
Title: Mi Puente: My Bridge to Better Cardiometabolic Health and Well-Being
Acronym: Mi Puente
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Principal Investigator, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01NR015754-01 (NIH)
Record Dates: First submitted 2015-12-01; First posted 2016-03-30 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes Mellitus; Cardiometabolic Conditions; Behavioral Health Concerns
Keywords: Hispanic Americans; Mental Health; Multimorbidity; Patient Readmission; Transitional Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Volunteer Peer Mentor + Behavioral Health Nurse
  Interventions: Behavioral: Volunteer Peer Mentor+Behavioral Health Nurse
- Control (No Intervention): Care as Usual

INTERVENTIONS:
Behavioral: Volunteer Peer Mentor+Behavioral Health Nurse — Intervention group participants receive intervention services from a Volunteer Peer Mentor and a Behavioral Health Nurse
  Other Names: Volunteer Peer Mentor (VPM) + Behavioral Health Nurse (BHN)
  Arms: Intervention Group

SUMMARY:
Mi Puente (or "My Bridge") is a culturally-tailored, interdisciplinary approach designed to support at-risk Hispanic patients and their caregivers pre- and post-hospital discharge as they navigate the multi-level barriers that contribute to inequities in health care access and use, and in turn, perpetuate disparities in cardiometabolic and behavioral health. Mi Puente utilizes a sustainable nurse + volunteer peer team-based model, bridging partnership between inpatient and outpatient care settings to meet the integrated (i.e., physical and behavioral) health needs of Hispanics who are hospitalized with multiple chronic cardiometabolic conditions and one or more behavioral health concern(s). Participants will be tested at Scripps Mercy Hospital - a large, non-profit, safety net hospital located in the US/Mexico border region of South San Diego County, California. The proposed randomized controlled trial will test Mi Puente versus Usual Care (evidence-based, best practice discharge procedures) in improving hospital utilization, patient-reported, and cost effectiveness outcomes. Electronic medical records (EMR) will be used to identify eligible patients and examine primary outcomes.

DETAILED DESCRIPTION:
This study targets disparities in cardiometabolic disease prevalence and outcomes, and the unmet behavioral health needs in the US Hispanic population. Differences in the quantity and quality of health care targeted to and received by members of the Hispanic population contribute to these disparities. Inequities in health care access and use are likely the result of an interaction of several multi-level factors, such as those related to low Socio-Economic Status (e.g., lack of transportation or health coverage, time constraints, unsafe environments, knowledge barriers), cultural factors, language or communication-style differences, and others. Mi Puente (or "My Bridge") is a culturally-tailored, interdisciplinary approach designed to support at-risk Hispanic patients and their caregivers pre- and post-hospital discharge as they navigate the multi-level barriers that contribute to inequities in health care access and use, and in turn, perpetuate disparities in cardiometabolic and behavioral health. Mi Puente builds upon a sustainable nurse + volunteer peer team-based model and a strong collaborative, bridging partnership between inpatient and outpatient care settings to meet the integrated (i.e., physical and behavioral) health needs of Hispanics who are hospitalized with multiple chronic cardiometabolic conditions and one or more behavioral health concern(s). The program is guided by the Social Ecological Model,34 Resources and Support for Self-Management Model,35,36 and Transtheoretical Model of behavior change,37,38 and will be tested at Scripps Mercy Hospital - a large, non-profit, safety net hospital located in the US/Mexico border region of South San Diego County, California. The proposed randomized controlled trial will test Mi Puente versus Usual Care (evidence-based, best practice discharge procedures) in improving hospital utilization, patient-reported, and cost effectiveness outcomes. Electronic medical records (EMR) will be used to identify eligible patients and examine primary outcomes. Ultimately the investigators seek to evaluate an effective, culturally appropriate, sustainable, and scalable program that addresses integrated health needs and reduces health disparities in Hispanics and other at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

1. Must be Hispanic
2. Must be ≥18 years
3. Must have ≥2 cardiometabolic conditions (e.g., obesity, diabetes, hypertension, dyslipidemia ischemic heart diseases, congestive heart failure, other chronic coronary conditions)
4. Must have ≥1 behavioral health concern(s) (i.e., related to mental health, life stressors, medication adherence, healthcare use)
5. Must have telephone access

Exclusion Criteria:

1. Pregnancy
2. Serious life-threatening condition with life expectancy < 6 months
3. Psychiatric morbidity or neurological/cognitive impairment of sufficient severity to preclude participation in the intervention
4. Discharging to location other than home (e.g., nursing care)
5. Does not speak Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute; Linda Gallo, PhD, Principal Investigator — San Diego State University
Locations (1):
- Scripps Mercy Chula Vista, Chula Vista, California, United States

REFERENCES:
- [Derived] Gallo LC, Fortmann AL, Clark TL, Roesch SC, Bravin JI, Spierling Bagsic SR, Sandoval H, Savin KL, Gilmer T, Talavera GA, Philis-Tsimikas A. Mi Puente (My Bridge) Care Transitions Program for Hispanic/Latino Adults with Multimorbidity: Results of a Randomized Controlled Trial. J Gen Intern Med. 2023 Jul;38(9):2098-2106. doi: 10.1007/s11606-022-08006-1. Epub 2023 Jan 25. PMID 36697929
- [Derived] Gallo LC, Fortmann AL, Bravin JI, Clark TL, Savin KL, Ledesma DL, Euyoque J, Sandoval H, Roesch SC, Gilmer T, Talavera GA, Philis-Tsimikas A. My Bridge (Mi Puente), a care transitions intervention for Hispanics/Latinos with multimorbidity and behavioral health concerns: protocol for a randomized controlled trial. Trials. 2020 Feb 12;21(1):174. doi: 10.1186/s13063-019-3722-8. PMID 32051005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2016 and March 2020, the study enrolled 536 inpatients of a hospital in South San Diego County that serves a mostly Hispanic/Latino, low socio-economic status patient population.
Pre-assignment Details: The target sample size based on power analysis was N=560. Enrollment was paused in March 2020, and then concluded early due to the COVID-19 pandemic. Because the design accommodated a 20% attrition rate, sample size was adequate for analysis of all outcomes.
Groups:
- Intervention Group: Volunteer Peer Mentor + Behavioral Health Nurse
  Volunteer Peer Mentor+Behavioral Hlth Nurse: Intervention group participants receive intervention services from a Volunteer Peer Mentor and a Behavioral Health Nurse
Period: Overall Study
Arm/Group | Intervention Group | Control
Started | 271 | 265
Completed | 186 | 175
Not Completed | 85 | 90
Not completed — Death | 17 | 13
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Lost to Follow-up | 57 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control | Total
Number analyzed (Participants) | 271 | 265 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.94 (14.10) | 62.66 (12.21) | 62.30 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 124 | 257
  Male | 138 | 141 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 271 | 265 | 536
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 1 | 3
  White | 83 | 67 | 150
  More than one race | 14 | 21 | 35
  Unknown or Not Reported | 166 | 171 | 337
Region of Enrollment [Number; unit: participants]
  United States | 271 | 265 | 536
Less than High School Education [Count of Participants; unit: Participants] | 113 | 134 | 247
Income Less than 30,000 per year [Count of Participants; unit: Participants] | 207 | 207 | 414
Not Employed [Count of Participants; unit: Participants] | 207 | 204 | 411
Married or Cohabitating [Count of Participants; unit: Participants] | 123 | 137 | 260
Born in Mexico [Count of Participants; unit: Participants] | 186 | 204 | 390
Primary Language is Spanish [Count of Participants; unit: Participants] | 200 | 212 | 412
Has Some Type of Health Insurance [Count of Participants; unit: Participants] | 248 | 247 | 495
Cardiometabolic Conditions [Mean (Standard Deviation); unit: cardiometabolic conditions] | 3.31 (1.33) | 3.35 (1.41) | 3.33 (1.37)
Behavioral Health Concerns [Mean (Standard Deviation); unit: behavioral health concerns] | 2.93 (1.56) | 3.03 (1.66) | 2.98 (1.61)
LACE Index -Length of Patient Stay in the Hospital, Acuity of Admission, Comorbidity, Emergency Vist [Mean (Standard Deviation); unit: LACE Index] — LACE index [a predictor of readmission and mortality risk that considers length of stay, admission acuity, comorbidities, and emergency department use, and ranges from 1 (lowest risk) to 19 (highest risk)].
  LACE Index | 7.26 (2.41) | 7.47 (4.45) | 7.36 (2.33)
Hospital Visit Length of Stay in Days [Mean (Standard Deviation); unit: days] | 4.87 (4.95) | 4.45 (5.52) | 4.66 (5.24)
Patient-Reported Outcomes Measurement Information System Global-10 Health Scale [Mean (Standard Deviation); unit: units on a scale] — This measure provides an overall score of self-reported physical and mental health.
  units on a scale | 26.91 (6.00) | 26.63 (6.23) | 26.8 (6.12)
Patient Activation Measure (PAM) - 13 Item [Mean (Standard Deviation); unit: units on a scale] | 60.14 (11.40) | 61.85 (12.33) | 60.99 (11.86)
Self-Management Resources for Chronic Disease, Chronic Illness Resources Survey (CRIS) [Mean (Standard Deviation); unit: units on a scale] | 2.80 (0.68) | 2.78 (0.63) | 2.79 (0.65)
Outpatient Visits Over the Past 3 Months [Mean (Standard Deviation); unit: outpatient visits] | 4.82 (7.20) | 4.42 (6.83) | 4.62 (7.01)
Urgent Care/Emergency Department Visits Over the Past 3 Months [Mean (Standard Deviation); unit: urgent care and ED visits] | 1.55 (1.73) | 1.49 (2.49) | 1.52 (2.11)
Inpatient Days Over the Past 3 Months [Mean (Standard Deviation); unit: inpatient days] | 4.47 (9.17) | 2.87 (5.33) | 3.67 (7.25)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least 1 Hospital Readmission Within 30 Days After Enrollment
Description: Number of patients with at least one hospital readmission within 30 days after enrollment
Time Frame: 30 days from baseline
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 271 | 265
participants | 43 | 25
Statistical Analysis 1: Comparison: Intervention Group vs Control; Analyzed using logistic regression analysis; Test type: Superiority; p = 0.01, Regression, Logistic

2. Primary Outcome: Number of Patients With at Least 1 Hospital Readmission Within 180 Days After Enrollment
Description: Number of patients with at least one hospital readmission within 180 days after enrollment
Time Frame: 180 days from baseline
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 271 | 265
participants | 120 | 98
Statistical Analysis 1: Comparison: Intervention Group vs Control; Test type: Superiority; p = 0.19, Regression, Logistic

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale - Patient-reported Outcome
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale - Patient-reported Outcome The minimum score on this scale is 10 and the maximum score on this scale is 50.
  A higher score on this scale means a better outcome. This measure provides an overall score of self-reported physical and mental health.
Time Frame: 6 months from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 271 | 265
score on a scale | 29.74 (7.32) | 29.57 (7.13)
Statistical Analysis 1: Comparison: Intervention Group vs Control; multilevel model analysis, random intercepts and slopes, appropriate link function for outcome, full maximum likelihood estimation; Test type: Superiority; p = 0.73, multilevel model analysis, random interc — P-value is for the time by group interaction effect, testing the difference in rate of change between the Intervention and Control groups from baseline to 6 months post baseline

4. Secondary Outcome: Patient Activation Measure (PAM) 13-Item - Patient-reported Outcome
Description: Patient Activation Measure (PAM) 13-Item - Patient-reported Outcome The minimum score for this scale is 0 and the maximum score for this scale is 100.
  A higher score on this scale is more patient activation and is a better outcome.
  This measure provides an overall score of patient activation.
Time Frame: 6 months from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 271 | 265
score on a scale | 66.15 (11.87) | 66.81 (14.45)
Statistical Analysis 1: Comparison: Intervention Group vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.28, multilevel model analysis, random interc — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Self-Management Resources for Chronic Disease, Chronic Illness Resources Survey (CIRS) - Short Version - Patient-reported Outcome
Description: Self-Management Resources for Chronic Disease, Chronic Illness Resources Survey (CIRS) - short version - patient-reported outcome The minimum score is 1 and the maximum score is 5. A higher score is a better outcome. This measure provides an overall score of support for healthful lifestyle behaviors and self-management from multiple sources.
Time Frame: 6 months from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 271 | 265
score on a scale | 3.14 (0.69) | 3.14 (0.68)
Statistical Analysis 1: Comparison: Intervention Group vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.71, multilevel model analysis, random interc — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Number of Outpatient Visits Over the Past 6 Months - Patient-reported
Description: Number of Outpatient Visits Over the Past 6 Months - Patient-reported - Outpatient Healthcare Utilization This measure assesses outpatient healthcare utilization by capturing the number of self-reported outpatient visits completed in the past 6 months. The minimum number of outpatient visits is 0. There is not set maximum. A higher score is a better outcome.
Time Frame: 6 months from baseline
Measure: Mean (Standard Deviation); unit: outpatient visits
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 271 | 265
outpatient visits | 5.39 (7.79) | 4.39 (6.79)
Statistical Analysis 1: Comparison: Intervention Group vs Control; negative binomial regression model analysis; Test type: Superiority; p = 0.42, negative binomial regression model analy

ADVERSE EVENTS:
Time Frame: 180 days
Description: All cause mortality
Arm/Group | Intervention Group | Control
All-Cause Mortality (participants affected / at risk) | 17/271 | 13/265
Serious Adverse Events (participants affected / at risk) | 0/271 | 0/265
Other Adverse Events (participants affected / at risk) | 0/271 | 0/265

LIMITATIONS AND CAVEATS:
The study may not have captured all readmissions since there are many regional hospitals. Other evolving approaches, such as the use of statewide health information exchanges, may improve ascertainment in future research. We did not delineate preventable from nonpreventable readmissions and did not have information on readmission acuity. Although some hospitalizations may have occurred due to COVID-19, it is likely that this affected both groups equally.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT02723019/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02723019/ICF_001.pdf